CLINICAL TRIAL: NCT01922726
Title: Registry of Sleep Apnea Monitoring and Atrial Fibrillation in Pacemaker Patients
Brief Title: Registry of Sleep Apnea Monitoring and Atrial Fibrillation in Pacemaker Patients (RESPIRE)
Status: Completed | Type: Observational
Sponsor: MicroPort CRM (Industry)
Responsible Party: Sponsor
Other Study IDs: RBSY03 - RESPIRE
Record Dates: First submitted 2013-08-01; First posted 2013-08-14 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Bradycardia
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to evaluate at 12 Months follow-up the association between Atrial Fibrillation (AF) and Sleep Apnea (SA) severity based on data measured and stored in REPLY 200 DR pacemaker.

DETAILED DESCRIPTION:
The object of the investigation relates to the function named Sleep Apnea Monitoring or SAM function. This function is part of the REPLY 200 DR pacemakers, whose intended use is cardiac pacing. Sleep Apnea Syndrom (SAS) causes serious social and economic problems, not only because of its high prevalence but also because it is associated with increased cardiovascular morbidity and mortality.

Patients with Sleep Apnea often have arterial and pulmonary hypertension, a high risk of coronary artery disease, and heart failure, whereas a high percentage of patients show heart rhythm disturbances. In addition, these patients are at increased risk of being involved in traffic accidents, as well as suffering a decline in their family, social, and professional lives. Therefore, the prompt diagnosis of these patients could be of great importance. Today the gold standard for the diagnosis of SAS is overnight polysomnography (PSG) in a sleep laboratory. However, the shortage of sleep laboratories and the high cost of PSG render this method inadequate for widespread screening. For these reasons, in recent years, there have been attempts to develop alternative diagnostic with a view to simplify the diagnosis.

Thanks to the feature SAM included in the pacemaker, sequences of respiratory cycles are analyzed to detect, to count and to report abnormal breathing events during the night. This analysis is based on the Minute Ventilation (MV) signal. The MV signal represents the real time expansion/contraction of the thorax of the patient. It is derived of the transthoracic impedance periodic measurements. The device is able to provide the physician with day-by-day Respiratory Disturbance Index (RDI) equal to the sum of events divided by the number of hours per night. Physician will also access to the total number of events over the previous night presented per hour.

ELIGIBILITY:
Inclusion Criteria:

* Patient eligible for implantation of a dual-chamber pacemaker according to current available guidelines
* Patient with REPLY 200 DR implantation performed
* Patient who provides signed and dated informed consent (according to the laws and regulations of the country in which the observational study is conducted)

Exclusion Criteria:

* Inability to understand the purpose of the study or refusal to co-operate
* Unavailability for routine follow-ups at the implanting centre
* Already included in another clinical study that could affect the results of this study
* Inability or refusal to provide informed consent
* Patient is minor (less than 18-years old)
* Patient is pregnant
* Patient is forfeiture of freedom or under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient eligible for implantation of a dual-chamber pacemaker (primo-implant, replacement, upgrade) according to current available guidelines Patient with REPLY 200 DR implantation performed. Patient who provides signed and dated informed consent according to the local laws and regulations
Sampling Method: Probability Sample
Enrollment: 1257 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2017-03-20 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluate at 12 Months follow-up the association between Atrial Fibrillation (AF) and Sleep Apnea (SA) severity based on data measured and stored in the pacemaker. | 12 months
  The primary endpoint is to prove that the difference in AF occurrence between severe SA patients versus non severe is greater or equal to 6 % after 12 Months follow-up. AF will be measured using the Fallback Mode Switch duration (FMS) and SA using the Respiratory Disturbance Index (RDI), both stored in the device.
Collect all major serious adverse events as reported by the investigator during the duration of the study corresponding to death, myocardial infarction, stroke and re- intervention. | 18 months
  The co-primary endpoint is to evaluate the rate of composite endpoint of all major serious adverse events as reported by the investigator over 18 months follow up corresponding to death, myocardial infarction, stroke and re-intervention (at least one of the 4 types of major SAE per patient). These major SAE will be also assessed by type.

SECONDARY OUTCOMES:
Assess prevalence of SA in pacemaker population based on RDI measured and stored in the pacemaker at 1, 6, 12 and 18 Months. | 1, 6, 12 and 18 months
  The prevalence of SA will be calculated considering the sum of SA patients out of all patients having performed the given follow up.
  Patients known as treated for SAS could not be taken into account in a secondary analysis.
Evaluate at 1, 6, 12 and 18 Months follow-up the association between subclinical atrial fibrillation and sleep apnea based on data measured and stored in the pacemaker. | 1, 6, 12 and 18 months
  Same method as described in outcome 1 except in this secondary objective, a patient will be considered as presenting subclinical AF when presenting between enrolment and a given follow up (M1, M6, M12 or M18) at least one fallback mode switch episode as following:
  * 1st case: below or equal to 6 minutes in the same day
  * 2nd case: between 6 minutes and 6 hours 17 in the same day
  * 3rd case: strictly greater than 6 hours17 in the same day.
Evaluate at 1, 6 and 18 Months follow-up the association between AF and SA severity based on data measured and stored in the pacemaker (qualitative data). | 1, 6 and 18 months
  The definition and method are the same as described in outcome 1 except measurements will be performed at 1, 6 and 18 Months.
Evaluate at 1, 6, 12 and 18 Months follow-up the association between AF and SA severity based on data measured and stored in the pacemaker (quantitative data). | 1, 6, 12 and 18 months
  Same method as described in outcome 1 except in this secondary objective, a patient will be considered as presenting AF based on the FMS burden value. FMS burden is the time spent in fallback mode switch divided by the follow up period in days. This FMS will be measured between 2 consecutives available follow up: enrolment and M1, then M1 and M6, M6 and M12, M12 and M18.
Evaluate at 1, 6, 12 and 18 Months follow-up the association between AF diagnosed on clinical assessment (ECG, holter, AF related serious adverse events: cardioversion, ablation…) and SA severity. | 1, 6, 12 and 18 months
  The AF episode diagnosed on clinical assessment will be collected in CRF at each follow up (M1, M6, M12 and M18). The RDI stored at the date of each AF event will be collected. We will then measure out of all AF events, how many of them are associated with a severe Sleep Apnea (RDI >=20).
Occurrence of patients referred to sleep specialists - Occurrence of patients referred to sleep specialists. - Occurrence of patients having sleep exam during the study. - Occurrence patients being treated for SA during the study. | 1, 6, 12 and 18 months
  The aim of this secondary objective was to observe how cardiologists in their routine practice would use this new information offered by SAM function (RDI). In particular, the physician process to decide whether he/she refers the patient to a sleep specialist will be observed. At each follow up the cardiologist asked the patient whether he/she had any visit to a sleep specialist since the last follow-up (pneumologist, neurologist, Ear Nose and Throat specialist …).
  For the patients evaluable at each of the scheduled visits, the number and percentage of patients who made a visit to a sleep specialist were to be presented overall and by the type of specialist (pneumologist, neurologist, Ear Nose and Throat specialist, etc) for severe and non-severe SA patients.
Occurrence of patients having sleep exam during the study | 1, 6, 12 and 18 months
  The aim of this secondary objective was to observe whether patients will undergo further sleep investigations (Polygraphy, Polysomnography…).
  At each follow up the cardiologist asked the patient whether he/she had any sleep exam since the last follow-up (Polygraphy, Polysomnography, oxymetry). Then the data was filled in the patient CRF.
  For the patients evaluable at each of the scheduled visits, the number and percentage of patients who underwent a sleep exam were to be presented overall and by the type of test (Polygraphy, Polysmonography, Oxymetry, etc).
Compare the sleep lab results with the RDI stored in the pacemaker | 1, 6, 12 and 18 months
  At each follow-up visit, the patients who did undergo aSleep Apnea test and were diagnosed as having SA were considered a patient with SA as per Lab results.
  The association of SA as diagnosed by Lab results with that of SA as measured based on RDI values were presented based on true positive/negative and false positive/negative.
Occurrence of patients being treated for SA during the study | 1, 6, 12 and 18 months
  At each follow up the cardiologist asked the patient whether he/she had any treatment for Sleep Apnea. Then the data was filled in the patient CRF. Then at each time-point, the number and percentages of evaluable patients who had been treated for SA will be presented by the definition of severe/non-severe SA
Compare RDI before and after SA treatment | 1, 6, 12 and 18 months
  The aim of this secondary objective was to assess how the SA treatment impacted the level of RDI stored in the device. It was observed in different studies that, to assess the benefit of SA treatments, a follow-up period of 4 to 16 weeks was recommended.
Compare AF (using FMS duration and AF related hospitalization) before and after SA treatment when the patient is treated | 1, 6, 12 and 18 months
  The aim of this secondary objective was to assess how SA treatment impacted the AF using FMS duration. It was observed in different studies that, to assess the benefit of SA treatments, a follow-up period of 4 to 16 weeks was recommended.
Stability of the RDI. | 1, 6, 12 and 18 months
  The RDI variability was determined with the measure of Standard Deviation calculated based on all the daily RDI values. The relationship between this measure of RDI variability with RDI, SA diagnosis and SA treatment will be assessed. A high value of SD indicated greater instability in daily RDI values compared to a lower SD.
Association between SA severity and indication for pacemaker's implantation. | 18 months
  The aim is to investigate the severity of SA according to the patient's pacing indications. The implant indication will be collected at enrollment and is described as II° AVB, III° AVB, Syncope, Brady-Tachy Syndrome, Sinus Node Dysfunction, Carotid Sinus Syndrome. For each implant indication, the number and percentages of severe and non-severe SA patients will be presented.
Collect serious adverse events throughout the study. | 1, 6, 12 and 18 months
  Serious adverse events will be collected to verify the absence of unanticipated adverse effects due to the device.
Evaluate at given time points any correlation between data stored in the device and clinical assessment related to the primary and secondary endpoints. | 1, 6, 12 and 18 months
  Evaluate at given time points any correlation between data stored in the device and clinical assessment related to the primary and secondary endpoints.

CONTACTS AND LOCATIONS:
Overall Officials: Julio MARTI ALMOR, Dr, Principal Investigator — Hospital Del Mar, Barcelona, Spain
Locations (1):
- Hospital Del Mar, Barcelona, Spain

REFERENCES:
- [Derived] Marti-Almor J, Marques P, Jesel L, Garcia R, Di Girolamo E, Locati F, Defaye P, Venables P, Dompnier A, Barcelo A, Nagele H, Burri H. Incidence of sleep apnea and association with atrial fibrillation in an unselected pacemaker population: Results of the observational RESPIRE study. Heart Rhythm. 2020 Feb;17(2):195-202. doi: 10.1016/j.hrthm.2019.09.001. Epub 2019 Sep 4. PMID 31493591